CLINICAL TRIAL: NCT00320528
Title: An Open-Label Study of the Efficacy of Atomoxetine Hydrochloride on Quality of Life of Children and Adolescents With Attention-Deficit/Hyperactivity Disorder With or Without Comorbid Conditions
Brief Title: Efficacy of Atomoxetine on Psychosocial Function of Children and Adolescents With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9867; B4Z-IT-LYDS
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Results first posted 2010-01-06 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2009-12

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pure ADHD (Experimental): Attention-Deficit/Hyperactivity Disorder (ADHD) alone. Received atomoxetine: 0.5 milligrams per kilogram per day (mg/kg/day), by mouth (PO) for 1 week then 1.2 mg/kg/day, PO for 11 weeks followed by up to 1.4 mg/kg/day, PO for up to 12 additional weeks
  Interventions: Drug: atomoxetine
- ADHD+Internalizing Disorders (Experimental): Attention-Deficit/Hyperactivity Disorder (ADHD) plus internalizing disorders. Received atomoxetine: 0.5 milligrams per kilogram per day (mg/kg/day), by mouth (PO) for 1 week then 1.2 mg/kg/day, PO for 11 weeks followed by up to 1.4 mg/kg/day, PO for up to 12 additional weeks
  Interventions: Drug: atomoxetine
- ADHD+Externalizing Disorders (Experimental): Attention-Deficit/Hyperactivity Disorder (ADHD) plus externalizing disorders. Received atomoxetine: 0.5 milligrams per kilogram per day (mg/kg/day), by mouth (PO) for 1 week then 1.2 mg/kg/day, PO for 11 weeks followed by up to 1.4 mg/kg/day, PO for up to 12 additional weeks
  Interventions: Drug: atomoxetine

INTERVENTIONS:
Drug: atomoxetine — 0.5 milligrams per kilogram per day (mg/kg/day), by mouth (PO) for 1 week then 1.2 mg/kg/day, PO for 11 weeks followed by up to 1.4 mg/kg/day, PO for up to 12 additional weeks
  Other Names: LY139603; Strattera

SUMMARY:
This study aims to assess the effectiveness of atomoxetine on psychosocial functioning and emotional well being of children and adolescents with ADHD and to evaluate whether and in what measure the presence of comorbid conditions (internalizing and externalizing disorders) influences atomoxetine's ability to improve the quality of life of ADHD subjects.

ELIGIBILITY:
Inclusion Criteria:

* Child or adolescent patients, male or female outpatients, who are at least 6 years of age, but must not yet have reached their 16th birthday prior to Visit 1, when informed consent is obtained
* Patients must meet Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) diagnostic criteria for ADHD (any subtype) and score at least 1.5 standard deviations above the age norm for their diagnostic subtype using published norms for the Swanson, Nolan and Pelham Questionnaire: Attention-Deficit/Hyperactivity Disorder Subscale (SNAP-IV ADHD Subscale) score at both Visit 1 and 2
* Laboratory results, including serum chemistries, hematology, and urinalysis, must show no clinically significant abnormalities (clinically significant is defined as laboratory values requiring acute medical intervention, indicating a serious medical illness, or requiring further medical evaluation in the judgment of the investigator)
* An electrocardiogram (ECG) must be performed to exclude cardiac diseases at the baseline/screening visit and the results must be reviewed by the investigator at Visit 2 prior to dispensing of study material
* Patients and parents have been judged by the investigator to be reliable to keep appointments for clinic visits and all tests, including venipuncture, and examinations required by the protocol.

Exclusion Criteria:

* Patients who have a documented history of Bipolar I or II disorder, any history of psychosis or pervasive development disorder
* Patients with a history of any seizure disorder (other than febrile seizures) or patients who have taken (or are currently taking) anticonvulsants for seizure control are not eligible to participate
* Patients at serious suicidal risk as assessed by the investigator
* Patients with significant cardiovascular disease or other conditions that could be aggravated by an increased heart rate or increased blood pressure
* Patients who have any medical condition that would increase sympathetic nervous system activity markedly (for example, catecholamine-secreting neural tumor), or who are taking a medication on a daily basis (for example, albuterol, inhalation aerosols, pseudoephedrine), that has sympathomimetic activity. Such medications can be taken on an as-needed basis

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 269 (Actual)
Dates: Start 2006-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (20):
- Italy (20):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Acireale
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Avellino
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bosisio Parini
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brescia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Catania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coppito
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cremona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ostuni
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palermo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Perugia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sassari
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Savigliano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Siena
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trieste
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Troina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Udine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Viterbo

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study Period I was a 3-day screening period. Study Period II was 12 weeks long. Study Period III was an optional additional 12 week open-label extension. Results are presented for Period II (patients who received at least one dose of study drug).
Period: Study Period II
Arm/Group | Pure ADHD | ADHD+Internalizing Disorders | ADHD+Externalizing Disorders
Started | 98 | 41 | 130
Received at Least One Dose of Study Drug | 97 | 38 | 128
Completed | 87 | 31 | 108
Not Completed | 11 | 10 | 22
Not completed — Adverse Event | 3 | 4 | 8
Not completed — Parent/Caregiver Decision | 8 | 3 | 11
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Entry Criteria Exclusion | 0 | 2 | 2
Period: Study Period III
Arm/Group | Pure ADHD | ADHD+Internalizing Disorders | ADHD+Externalizing Disorders
Started | 87 | 31 | 108
Completed | 0 | 0 | 2
Not Completed | 87 | 31 | 106
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 2
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Parent/Caregiver Decision | 14 | 3 | 11
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 2
Not completed — Sponsor Decision | 0 | 0 | 1
Not completed — Atomoxetine Commercially Available | 68 | 25 | 90

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pure ADHD | ADHD+Internalizing Disorders | ADHD+Externalizing Disorders | Total
Number analyzed (Participants) | 97 | 38 | 128 | 263
Age Continuous [Mean (Standard Deviation); unit: years] | 10.12 (2.51) | 10.42 (2.41) | 10.00 (2.57) | 10.11 (2.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 3 | 9 | 26
  Male | 83 | 35 | 119 | 237
Region of Enrollment [Number; unit: participants]
  Italy | 97 | 38 | 128 | 263
Race/Ethnicity [Number; unit: participants]
  Caucasian | 90 | 36 | 124 | 250
  Hispanic | 1 | 2 | 2 | 5
  African | 3 | 0 | 0 | 3
  Native American | 1 | 0 | 2 | 3
  East Asian | 2 | 0 | 0 | 2
Child Health and Illness Profile - Child Edition (CHIP-CE) - Achievement Domain [Mean (Standard Deviation); unit: T-Score] — Parent-rated assessment of a child's health status and level of functioning. It consists of 76 items. The majority of items assess frequency of activities or feelings using a five-point response format (for example, 'how good is your child at making friends?' 1=never, 5=always). Standard scores (t-value) were established, with all domains and subdomains having a mean score of 50 and standard deviation of 10. Standard scores are expressed in standard deviation units. Achievement Domain Range = -3.1 to 67.7. Higher scores mean greater health or level of functioning in achievement.
  T-Score
    Achievement Domain (N=96, N=33, N=121) | 29.27 (7.89) | 27.72 (7.73) | 25.83 (7.60) | 27.40 (7.86)
    Satisfaction Domain (N=96, N=24, N=122) | 39.26 (13.89) | 30.11 (14.83) | 31.69 (14.78) | 34.34 (14.91)
    Comfort Domain (N=96, N=35, N=122) | 51.31 (9.40) | 46.76 (12.28) | 44.74 (9.38) | 47.51 (10.26)
    Resilience Domain (N=96, N=34, N=123) | 39.34 (10.15) | 34.96 (10.89) | 31.40 (11.85) | 34.89 (11.65)
    Risk Avoidance (N=96, N=33, N=121) | 32.03 (9.7) | 30.48 (12.29) | 22.85 (12.00) | 27.38 (12.01)
Children's Depression Rating Scale-Revised (CDRS-R) [Mean (Standard Deviation); unit: units on a scale] — Measures presence and severity of depression. Consists of 17 items scored on a 1-5 or 1-7 scale. A rating of 1 indicates normal, thus the minimum score is 17. The maximum score is 113. In general, scores below 20 indicate an absence of depression; scores of 20 or 30 indicate borderline depression; scores of 40 to 60 indicate moderate depression.
  units on a scale | 37.93 (12.26) | 43.76 (13.48) | 43.06 (13.69) | 41.26 (13.35)
Clinical Global Impression-Attention Deficit Hyperactivity Disorder-Severity Scale (CGI-ADHD-S) [Mean (Standard Deviation); unit: units on a scale] — Measures severity of the patient's overall severity of ADHD symptoms (1=normal, not at all ill; 7=among the most extremely ill patients).
  units on a scale | 4.64 (0.79) | 4.97 (0.79) | 4.98 (0.78) | 4.85 (0.80)
Conners' Teacher Rating Scale-Revised:Short Form (CTRS-R:S) [Mean (Standard Deviation); unit: units on a scale] — A 28-item rating scale (0 [not at all/never] to 3 [very much true/very often]) completed by the teacher to assess problem behaviors related to ADHD. Subscale total scores range from 0 to 15 for Oppositional and Cognitive Problems, 0 to 21 for Hyperactivity, and 0 to 36 for ADHD Index.
  units on a scale
    Oppositional | 5.97 (4.93) | 4.97 (4.66) | 8.62 (4.83) | 7.10 (5.05)
    Cognitive Problems | 7.86 (3.73) | 7.68 (3.80) | 7.96 (3.61) | 7.88 (3.67)
    Hyperactivity | 11.38 (6.09) | 12.03 (5.21) | 14.67 (5.15) | 13.05 (5.74)
    ADHD Index | 22.14 (6.86) | 22.94 (6.01) | 25.18 (6.07) | 23.70 (6.52)
Pediatric Anxiety Rating Scale (PARS) [Mean (Standard Deviation); unit: units on a scale] — The Pediatric Anxiety Rating Scale (PARS) is used to rate the severity of anxiety in children and adolescents, ages 6 to 17 years. The total score for the PARS is derived by summing 5 of the 7 severity/impairment/interference items (2,3,5,6,7). The total score ranges from 0 (none) to 25 (extreme severity). Items 1 (overall number of anxiety symptoms) and 4 (overall severity of physical symptoms) are not included in the total score calculation.
  units on a scale | 2.50 (2.67) | 7.50 (5.68) | 4.67 (5.12) | 4.28 (4.76)
Swanson, Nolan, and Pelham Rating Scale Revised (SNAP-IV) [Mean (Standard Deviation); unit: units on a scale] — The SNAP-IV is a 26-item scale that includes 1 item for each of the 18 symptoms contained in the DSM-IV diagnosis of ADHD and 1 item for each of the 8 symptoms contained in the DSM-IV diagnosis of ODD. Each item is score on 0 to 3 scale (0 = "Not at All", 1 = "Just a Little", 2 = "Pretty Much", 3 = "Very Much"). The SNAP-IV yields scores in three domains: Inattention (items 1-9: subscore range=0-27), Hyperactivity/impulsivity (items 10-18: subscale range=0-27), and Oppositional (items 19-26: subscale range=0-24). Combined type (inattention + hyperactivity/impulsivity) scores range from 0-54.
  units on a scale
    Inattention Subscale (N=97, N=38, N=127) | 20.28 (4.19) | 21.03 (3.72) | 21.87 (3.48) | 21.16 (3.85)
    Hyperactivity/Impulsivity Subscale (N=97, N=38, N= | 17.21 (6.10) | 19.66 (5.54) | 21.04 (3.48) | 19.42 (5.19)
    Combined Type Subscale (N=97, N=38, N=127) | 37.48 (7.78) | 40.68 (7.87) | 42.91 (5.51) | 40.58 (7.20)
    Oppositional Subscale (N=97, N=38, N=127) | 10.15 (4.54) | 12.32 (4.67) | 17.99 (3.57) | 14.27 (5.51)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 12 Week Endpoint in Child Health and Illness Profile - Child Edition (CHIP-CE), Achievement Domain
Description: Parent-rated assessment of a child's health status and level of functioning. It consists of 76 items. The majority of items assess frequency of activities or feelings using a five-point response format (for example, 'how good is your child at making friends?' 1=never, 5=always). Standard scores (t-value) were established, with all domains and subdomains having a mean score of 50 and standard deviation of 10. Standard scores are expressed in standard deviation units. Achievement Domain Range = -3.1 to 67.7. Higher scores mean greater health or level of functioning in achievement.
Time Frame: Baseline, 12 Weeks
Population: Number of patients with baseline and at least one nonmissing post-baseline measurement.
Measure: Mean (95% Confidence Interval); unit: T-Score
Arm/Group | Pure ADHD | ADHD+Internalizing Disorders | ADHD+Externalizing Disorders
Number analyzed (Participants) | 83 | 28 | 97
T-Score | 2.65 [0.93 to 4.37] | 0.51 [-1.38 to 2.39] | 3.89 [2.22 to 5.57]

2. Secondary Outcome: Change From Baseline to 12 Week Endpoint in the Attention-Deficit/Hyperactivity Disorder (ADHD) Subscales of 18-Item Swanson, Nolan and Pelham Rating Scale (SNAP-IV)
Description: Items from the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) criteria for ADHD are included for the two subsets of symptoms: inattention (items #1-#9: total score=0-27) and hyperactivity/impulsivity (items #11-#19: total score=0-27). The SNAP-IV is based on a 0 (not at all) to 3 (very much) rating scale. Total combined type (inattention plus hyperactivity/impulsivity) subscale scores range from 0 to 54.
Time Frame: Baseline, 12 Weeks
Population: Number of patients with baseline and at least one nonmissing post-baseline measurement.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pure ADHD | ADHD+Internalizing Disorders | ADHD+Externalizing Disorders
Number analyzed (Participants) | 90 | 33 | 111
units on a scale
  Inattention Subscale | -5.88 [-6.97 to -4.78] | -5.52 [-7.34 to -3.69] | -7.58 [-8.69 to -6.46]
  Hyperactivity/Impulsivity Subscale | -6.19 [-7.25 to -5.13] | -5.67 [-7.41 to -3.92] | -8.08 [-9.09 to -7.07]
  Combined Type (ADHD) Subscale | -12.1 [-13.9 to -10.3] | -11.2 [-14.4 to -7.92] | -15.7 [-17.6 to -13.7]

3. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Clinical Global Impressions-ADHD-Severity (CGI-ADHD-S)
Description: Measures severity of the patient's overall severity of ADHD symptoms (1=normal, not at all ill; 7=among the most extremely ill patients).
Time Frame: Baseline, 12 Weeks
Population: Number of patients with baseline and at least one nonmissing post-baseline measurement.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pure ADHD | ADHD+Internalizing Disorders | ADHD+Externalizing Disorders
Number analyzed (Participants) | 88 | 32 | 112
units on a scale | -1.23 [-1.46 to -0.99] | -1.63 [-1.99 to -1.26] | -1.42 [-1.63 to -1.21]

4. Secondary Outcome: Change From Baseline to 12 Week Endpoint in CHIP-CE Satisfaction, Comfort, Resilience and Risk Avoidance Domains
Description: Parent-rated assessment of a child's health status and level of functioning. It consists of 76 items. The majority of items assess frequency of activities or feelings using a five-point response format (for example, 'how good is your child at making friends?' 1=never, 5=always). Standard scores (t-value) were established, with all domains having a mean score of 50 and standard deviation of 10. Satisfaction range=-25.7 to 66.3; Comfort=-28.6 to 67.2; Resilience=-36.3 to 71.8; Risk Avoidance=-23.5 to 62.5. Higher scores mean greater health or level of functioning in that domain.
Time Frame: Baseline, 12 Weeks
Population: Number of patients with baseline and at least one nonmissing post-baseline measurement.
Measure: Mean (95% Confidence Interval); unit: T-Score
Arm/Group | Pure ADHD | ADHD+Internalizing Disorders | ADHD+Externalizing Disorders
Number analyzed (Participants) | 97 | 38 | 128
T-Score
  Satisfaction Domain (N=88, N=31, N=105) | 2.14 [-0.06 to 4.34] | 0.81 [-3.33 to 4.95] | 3.78 [1.18 to 6.39]
  Comfort Domain (N=86, N=28, N=103) | 1.01 [-0.88 to 2.90] | 5.72 [1.24 to 10.19] | 4.94 [3.14 to 6.73]
  Resilience Domain (N=87, N=30, N=106) | 1.21 [-0.85 to 3.27] | 2.18 [-1.31 to 5.67] | 3.07 [1.10 to 5.03]
  Risk Avoidance Domain (N=82, N=28, N=94) | 4.72 [2.93 to 6.51] | 5.70 [1.96 to 9.45] | 9.88 [7.88 to 11.88]

5. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Pediatric Anxiety Rating Scale (PARS)
Description: The Pediatric Anxiety Rating Scale (PARS) is used to rate the severity of anxiety in children and adolescents, ages 6 to 17 years. The total score for the PARS is derived by summing 5 of the 7 severity/impairment/interference items (2,3,5,6,7). The total score ranges from 0 (none) to 25 (extreme severity). Items 1 (overall number of anxiety symptoms) and 4 (overall severity of physical symptoms) are not included in the total score calculation.
Time Frame: Baseline, 12 Weeks
Population: Number of patients with baseline and at least one nonmissing post-baseline measurement.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pure ADHD | ADHD+Internalizing Disorders | ADHD+Externalizing Disorders
Number analyzed (Participants) | 89 | 33 | 112
units on a scale | -0.18 [-0.70 to 0.34] | -1.88 [-3.40 to -0.36] | -1.18 [-1.90 to -0.46]

6. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Children's Depression Rating Scale-Revised (CDRS-R)
Description: Measures presence and severity of depression. Consists of 17 items scored on a 1-5 or 1-7 scale. A rating of 1 indicates normal, thus the minimum score is 17. The maximum score is 113. In general, scores below 20 indicate an absence of depression; scores of 20 or 30 indicate borderline depression; scores of 40 to 60 indicate moderate depression.
Time Frame: Baseline, 12 Weeks
Population: Number of patients with baseline and at least one nonmissing post-baseline measurement.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pure ADHD | ADHD+Internalizing Disorders | ADHD+Externalizing Disorders
Number analyzed (Participants) | 97 | 38 | 128
units on a scale | -1.60 [-3.54 to 0.34] | -2.56 [-6.38 to 1.25] | -3.13 [-4.64 to -1.62]

7. Secondary Outcome: Change From Baseline to 12 Week Endpoint in SNAP-IV Oppositional Scale
Description: Items are included from the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) criteria for Oppositional Defiant Disorder. The SNAP-IV is based on a 0 (not at all) to 3 (very much) rating scale. Total subscale scores range from 0 to 24.
Time Frame: Baseline, 12 Weeks
Population: Number of patients with baseline and at least one nonmissing post-baseline measurement.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pure ADHD | ADHD+Internalizing Disorders | ADHD+Externalizing Disorders
Number analyzed (Participants) | 90 | 33 | 111
units on a scale | -2.01 [-2.86 to -1.16] | -2.12 [-3.95 to -0.29] | -5.54 [-6.43 to -4.65]

8. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Adolescent Symptom Inventory-4: Parent Checklist (ASI-4)
Description: Parent-completed ASI-4 contains 120 items on 18 emotional and behavioral disorders in adolescents (12-18 years old). Item score range:0 (no symptoms) to 3 (maximum impairment). Categories: A=ADHD (0-54); B=Conduct (0-60); C=Oppositional Defiant (0-24); D=Generalized Anxiety (0-18); E=Specific Phobia/Panic Attack/Obsessions/Compulsions/Somatization (0-30); F=Social Phobia (0-6); G=Separation Anxiety (0-24); H=Schizoid Personality (0-9); I=Schizophrenia (0-6); J=Enuresis (0-18); K=Major Depressive (0-42); L=Bipolar (0-27); M=Anorexia (0-12); N=Bulimia (0-12); O=Substance Abuse (0-18).
Time Frame: Baseline, 12 Weeks
Population: Number of adolescent patients with baseline and at least one nonmissing post-baseline measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pure ADHD | ADHD+Internalizing Disorders | ADHD+Externalizing Disorders
Number analyzed (Participants) | 26 | 10 | 30
units on a scale
  Category A - Baseline | 32.73 (11.42) | 38.33 (10.32) | 38.13 (8.30)
  Category A - Change from Baseline | -11.4 (9.88) | -10.4 (11.55) | -11.6 (9.50)
  Category B - Baseline | 4.04 (4.25) | 6.00 (5.62) | 10.80 (5.41)
  Category B - Change from Baseline | -0.73 (2.92) | -0.60 (5.83) | -5.57 (5.58)
  Category C- Baseline | 7.92 (4.77) | 10.50 (3.72) | 15.60 (5.24)
  Category C - Change from Baseline | -0.88 (3.85) | -1.40 (6.15) | -5.47 (5.51)
  Category D- Baseline | 4.73 (3.14) | 9.20 (3.58) | 8.37 (3.54)
  Category D - Change from Baseline | -0.58 (3.09) | -1.70 (3.65) | -2.97 (3.67)
  Category E- Baseline | 3.58 (4.00) | 7.60 (7.85) | 3.63 (3.16)
  Category E - Change from Baseline | -0.38 (4.01) | -4.50 (8.72) | -1.30 (2.35)
  Category F- Baseline | 1.19 (1.27) | 2.60 (1.43) | 1.20 (1.37)
  Category F - Change from Baseline | -0.58 (0.81) | -1.40 (1.43) | -0.53 (1.25)
  Category G- Baseline | 2.27 (3.50) | 4.50 (5.25) | 2.10 (2.63)
  Category G - Change from Baseline | -0.46 (2.49) | -3.20 (4.71) | -0.97 (2.40)
  Category H- Baseline | 0.73 (1.28) | 1.60 (2.27) | 1.70 (1.74)
  Category H - Change from Baseline | -0.38 (1.20) | 0.20 (2.86) | -0.67 (1.69)
  Category I- Baseline | 1.00 (1.92) | 3.20 (3.65) | 2.13 (2.22)
  Category I - Change from Baseline | -0.19 (0.80) | -1.30 (3.89) | -0.93 (1.70)
  Category J- Baseline | 0.42 (0.99) | 0.40 (0.97) | 0.50 (0.78)
  Category J - Change from Baseline | 0.00 (0.69) | -0.30 (0.67) | -0.23 (0.43)
  Category K- Baseline | 3.73 (3.99) | 4.90 (2.85) | 4.23 (4.05)
  Category K - Change from Baseline | -1.04 (2.90) | -1.00 (3.50) | -1.60 (3.50)
  Category L- Baseline | 3.54 (4.68) | 5.10 (5.00) | 6.03 (5.02)
  Category L - Change from Baseline | -1.08 (3.46) | -0.20 (6.03) | -1.97 (4.30)
  Category M- Baseline | 0.73 (1.22) | 1.30 (2.06) | 0.50 (1.41)
  Category M - Change from Baseline | 0.15 (1.08) | -0.10 (3.21) | 0.30 (1.39)
  Category N- Baseline | 1.31 (1.54) | 2.20 (3.05) | 2.30 (1.84)
  Category N - Change from Baseline | -0.38 (1.70) | -0.90 (2.23) | -0.80 (1.49)
  Category O- Baseline | 0.23 (0.71) | 0.30 (0.95) | 0.53 (0.97)
  Category O - Change from Baseline | 0.15 (0.37) | -0.20 (0.63) | -0.13 (0.51)

9. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Child Symptom Inventory-4: Parent Checklist (CSI-4)
Description: The CSI-4 contains 97 items that screen for 15 emotional and behavioral disorders in children between 5 and 12 years old. Item score range:0 (no symptoms) to 3 (maximum impairment). Categories: A=ADHD (0-54); B=Conduct (0-60); C=Oppositional Defiant (0-24); D=Generalized Anxiety (0-18); E=Specific Phobia/Panic Attack/Obsessions/Compulsions/Somatization (0-30); F=Social Phobia (0-6); G=Separation Anxiety (0-24); H=Schizoid Personality (0-9); I=Schizophrenia (0-6); J=Enuresis (0-18).
Time Frame: Baseline, 12 Weeks
Population: Number of child patients with baseline and at least one nonmissing post-baseline measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pure ADHD | ADHD+Internalizing Disorders | ADHD+Externalizing Disorders
Number analyzed (Participants) | 58 | 22 | 78
units on a scale
  Category A - Baseline | 34.00 (10.43) | 36.00 (9.32) | 38.95 (8.68)
  Category A - Change from Baseline | -10.6 (9.76) | -9.68 (9.54) | -12.7 (12.06)
  Category B - Baseline | 9.29 (4.72) | 11.05 (4.13) | 15.65 (4.40)
  Category B - Change from Baseline | -2.12 (3.88) | -1.14 (5.25) | -3.76 (5.56)
  Category C - Baseline | 2.10 (2.44) | 2.23 (2.25) | 4.63 (3.69)
  Category C - Change from Baseline | -0.88 (2.11) | -0.05 (3.06) | -1.99 (3.17)
  Category D - Baseline | 5.83 (3.37) | 8.23 (3.96) | 7.41 (3.94)
  Category D - Change from Baseline | -0.84 (3.16) | -2.23 (3.01) | -1.63 (3.86)
  Category E - Baseline | 2.07 (1.87) | 2.09 (1.95) | 2.79 (2.69)
  Category E - Change from Baseline | -0.38 (1.90) | -0.41 (1.74) | -0.85 (2.43)
  Category F - Baseline | 0.48 (0.86) | 0.32 (0.57) | 0.91 (1.35)
  Category F - Change from Baseline | -0.17 (0.94) | -0.14 (0.64) | -0.24 (1.28)
  Category G - Baseline | 3.02 (2.70) | 4.05 (2.79) | 3.51 (3.30)
  Category G - Change from Baseline | -0.62 (2.40) | -0.91 (2.00) | -0.46 (2.52)
  Category H - Baseline | 3.66 (4.14) | 4.64 (4.02) | 4.45 (4.39)
  Category H - Change from Baseline | -1.10 (2.21) | -1.09 (2.93) | -1.54 (4.31)
  Category I - Baseline | 2.76 (1.85) | 2.77 (1.38) | 2.94 (1.93)
  Category I - Change from Baseline | -0.03 (1.83) | -0.45 (1.47) | -0.32 (1.75)
  Category J - Baseline | 3.92 (3.98) | 5.58 (6.05) | 5.22 (4.47)
  Category J - Change from Baseline | -1.34 (3.64) | -0.86 (2.61) | -1.55 (4.34)

10. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Conners' Teacher Rating Scale-Revised: Short Form (CTRS-R:S)
Description: A 28-item rating scale (0 [not at all/never] to 3 [very much true/very often]) completed by the teacher to assess problem behaviors related to ADHD. Subscale total scores range from 0 to 15 for Oppositional and Cognitive Problems, 0 to 21 for Hyperactivity, and 0 to 36 for ADHD Index.
Time Frame: Baseline, 12 Weeks
Population: Number of patients with baseline and at least one nonmissing post-baseline measurement.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pure ADHD | ADHD+Internalizing Disorders | ADHD+Externalizing Disorders
Number analyzed (Participants) | 60 | 15 | 53
units on a scale
  Oppositional | -1.42 [-2.22 to -0.61] | 1.07 [-0.33 to 2.46] | -2.35 [-3.55 to -1.15]
  Cognitive Problems | -1.08 [-1.72 to -0.45] | -0.47 [-1.74 to 0.80] | -0.94 [-1.77 to -0.11]
  Hyperactivity | -2.87 [-4.04 to -1.69] | -2.34 [-4.80 to 0.11] | -4.09 [-5.52 to -2.67]
  ADHD Index | -4.94 [-6.36 to -3.52] | -3.60 [-6.65 to -0.55] | -6.62 [-8.59 to -4.65]

ADVERSE EVENTS:
Arm/Group | Pure ADHD | ADHD+Internalizing Disorders | ADHD+Externalizing Disorders
Serious Adverse Events (participants affected / at risk) | 1/97 | 0/38 | 2/128
Other Adverse Events (participants affected / at risk) | 76/97 | 29/38 | 94/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pure ADHD (N=97) | ADHD+Internalizing Disorders (N=38) | ADHD+Externalizing Disorders (N=128)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Idiosyncratic drug reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pure ADHD (N=97) | ADHD+Internalizing Disorders (N=38) | ADHD+Externalizing Disorders (N=128)
Abdominal pain (Gastrointestinal disorders) | 9 (13) | 8 (9) | 18 (32)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 6 (8) | 12 (17)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (3) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 12 (17) | 10 (19) | 26 (36)
Vomiting (Gastrointestinal disorders) | 13 (23) | 6 (13) | 15 (20)
Asthenia (General disorders) | 5 (6) | 6 (6) | 7 (7)
Fatigue (General disorders) | 5 (5) | 0 (0) | 2 (3)
Irritability (General disorders) | 4 (4) | 6 (6) | 12 (16)
Pyrexia (General disorders) | 3 (3) | 0 (0) | 8 (8)
Gastroenteritis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 11 (15) | 1 (1) | 12 (15)
Anorexia (Metabolism and nutrition disorders) | 24 (26) | 11 (15) | 33 (39)
Decreased appetite (Metabolism and nutrition disorders) | 11 (13) | 7 (7) | 14 (20)
Headache (Nervous system disorders) | 20 (34) | 10 (17) | 26 (35)
Somnolence (Nervous system disorders) | 22 (23) | 11 (15) | 34 (44)
Aggression (Psychiatric disorders) | 4 (5) | 1 (1) | 9 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 8 (10)

LIMITATIONS AND CAVEATS:
The original intent was to also calculate change and 95% confidence intervals at end of Period III; however, due to low number of patients completing Period III, variations from baseline (LOCF), are not suitable for further analysis or description.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days